CLINICAL TRIAL: NCT02743754
Title: Hyperbaric Oxygen Therapy for Cardiac Surgery-Associated Acute Kidney Injury: A First-in-Human Pilot Study
Brief Title: Hyperbaric Oxygen Therapy and Acute Kidney Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-9843
Record Dates: First submitted 2015-11-30; First posted 2016-04-19 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Standard of Care; Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Therapy (Placebo Comparator): Standard supportive therapies for Acute Kidney Injury (AKI), which entail optimization of hemodynamics and hemoglobin levels.
  Interventions: Other: Standard therapy
- Standard Therapy and hyperbaric oxygen (Active Comparator): Standard therapies and treated in the hyperbaric chamber within 12 hours of surgery. There will be 4 hyperbaric oxygen treatments in 48 hours (1 every 12 hours), each treatment will last 90 minutes with 100% oxygen at 2.4 atmospheres absolute (ATA).
  Interventions: Other: Standard therapy; Other: Hyperbaric Oxygen

INTERVENTIONS:
Other: Standard therapy — The standard of care for improving oxygen delivery to the kidney. These may include blood transfusions for anemia, treatment of low blood pressure and oxygen for low blood oxygen levels.
Other: Hyperbaric Oxygen — The standard of care therapies and in addition will be treated in the hyperbaric chamber within 12 hours of surgery. There will be 4 hyperbaric oxygen treatments in 48 hours (1 every 12 hours), each treatment will last 90 minutes with 100% oxygen at 2.4 ATA.
  Arms: Standard Therapy and hyperbaric oxygen

SUMMARY:
Kidney injury is a serious complication of cardiac surgery that occurs in up to 30% of patients and increases the risk of adverse outcomes. Kidney injury initiates when oxygen supply to the kidney drops below levels that are needed for normal cellular function, causing tissue oxygen deficiency (hypoxia), activation of the inflammatory cascade, and oxidative stress. Together, these events further impair tissue oxygenation, culminating in impaired kidney function due to cellular injury and death.

There are no effective therapies for kidney injury after cardiac surgery, but there is evidence that recovery is possible if the processes of injury - i.e., impaired oxygen delivery, increased inflammatory response, and oxidative stress - are ameliorated soon after the onset of injury. Hyperbaric oxygen therapy (HBOT) - which entails the intermittent inhalation of 100% oxygen in a hyperbaric chamber at a pressure higher than one absolute atmosphere (> 760 mmHg) - has been shown to positively affect all of these processes (i.e., to improve tissue oxygenation, reduce inflammation, and reduce oxidative stress). Thus, we hypothesized that HBOT will reduce the severity of kidney injury after cardiac surgery if it is initiated soon after onset of injury. This hypothesis has not been tested in humans, but is supported by animal studies.

In this first-in-human, unblinded, controlled pilot trial, 20 adult patients who develop severe kidney injury soon after cardiac surgery will be randomized (after obtaining informed consent from the patient or surrogate) to standard-of-care or early HBOT. Severe kidney injury will be defined as a ≥30% drop in kidney function within 6 hours of surgery (as determined by change in creatinine from before surgery to Intensive Care Unit (ICU) admission). This degree of injury occurs in ~ 2% of patients and is associated with a 12-fold increase in the risk of complete kidney failure (requiring dialysis) or death. Patients will be excluded if they have any relative or absolute contraindications to HBOT (e.g., severe ventricular dysfunction, ventricular assist device, severe respiratory dysfunction, pneumothorax, bronchospasm).

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* any cardiac surgery with cardiopulmonary bypass surgery
* ≥30% drop in kidney function within 6 hours of surgery (determined by change in creatinine from before surgery to ICU admission)

Exclusion Criteria:

* Pre-existing renal dysfunction (creatinine > 177 µmol/L)
* claustrophobia
* seizure disorder
* severe respiratory dysfunction (PaO2/fraction of inspired oxygen (FiO2) ratio <150 on 100% O2 and Peep of 10)
* active asthma or bronchospasm
* severe chronic obstructive pulmonary disease
* history of spontaneous pneumothorax or untreated pneumothorax
* congestive heart failure with left ventricular ejection fraction < 30%
* evidence of ongoing myocardial ischemia
* presence of ventricular assist device or intra-aortic balloon pump
* chronic sinusitis
* chronic/ acute otitis media or major ear drum trauma
* current treatment with bleomycin, cisplatin, doxorubicin and disulfiram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention | 7 days
  The proportion of patients qualified but not consented and the proportion of patients completing the study from each group.
Safety of the intervention as assessed by adverse events | 7 days
  Adverse events that are related to the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Karkouti, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hopsital University Health Network, Toronto, Ontario, Canada